CLINICAL TRIAL: NCT06132373
Title: Assessing Implementation of Delivering Community-based, Peer-led Interventions for Mental Health Problems Among Youth in Eldoret, Kenya
Acronym: Husisha
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Moi Teaching and Referral Hospital (Other); Academic Model Providing Access to Healthcare (AMPATH) (Other)
Responsible Party: Principal Investigator, Matthew Turissini, Assistant Professor of Clinical Medicine, Department of Medicine, Indiana University School of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: INTM-IIR-HUSISHA
Record Dates: First submitted 2023-11-01; First posted 2023-11-15 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2024-05

CONDITIONS: Unspecified Behavioral and Emotional Disorders With Onset Usually Occurring in Childhood and Adolescence; Mental Disorder First Evident in Infancy, Childhood, or Adolescence; Mental Disorder of Infancy, Childhood, or Adolescence (Diagnosis)
Keywords: Problem-solving therapy; Community Mental Health Services; Adolescents; Kenya
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: We will conduct a mixed-methods evaluation with peer providers, participants, and key delivery stakeholders such as FHOK staff. We will collect quantitative data from: (1) peer mentors prior to their training and during the delivery of screening and treatment, (2) participants prior to entering treatment and after treatment. We will track rates of retention, engagement, and attrition during screening and treatment delivery. Lastly, we will collect qualitative data including interviews with 10 purposively sampled participants and Focus Groups with peer mentors and key delivery stakeholders post-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm study (Experimental): We will apply evidence-based Problem Solving Therapy (PST), a transdiagnostic, low-intensity approach shown to improve mental health problems among adolescents with demonstrated effectiveness in global settings. PST for adolescents is a brief 5 session individual treatment with demonstrated efficacy when delivered by lay providers. PST is theorized to function by increasing adolescent capacity to cope with perceived and experienced stress through the use of problem- and emotion- focused coping skills that then allow engagement in positive, healthy activities.
  Interventions: Behavioral: Peer delivered problem solving therapy

INTERVENTIONS:
Behavioral: Peer delivered problem solving therapy — PST uses a straightforward approach amenable to use in new settings given its focus on idiographic problems, therefore session content is driven by the adolescent's presenting problem causing the most distress or impairment. We will use the standardized, core steps of PST and existing manualized protocols including from the Friendship Bench study and the WHO protocol for Problem Management Plus. The peers will deliver PST through 5 structured counseling sessions of 30-60 minutes over a 4-6 week period. There are 5 core components of PST which including problem listing and identification, problem exploration, developing an action plan, implementation, and follow up. The components will be introduced in the first session and be reviewed in an iterative process across the session to help participants use this model for different problems.

SUMMARY:
Introduction: Mental health disorders are a leading cause of disability among youth globally, and this has been worsened by the COVID-19 pandemic. In low and middle-income countries like Kenya and in rural Indiana, there is an enormous treatment gap for youth mental disorders due to limited mental health care resources.

Goals: The purpose of this project is to examine the implementation of community-based, peer-led management of mental health care screening, and treatment for adolescents in Eldoret, Kenya using the REAIM framework.

Methods: We shall conduct a one-week training to peer-mentors on screening for common mental health problems using the SDQ, PHQ-9, GAD-7, and YTP and treating adolescents who screen positive using a 5 session Problem Solving Treatment (PST), an evidence-based treatment for common youth mental health problems. We will then select five of the peers to deliver the intervention under the supervision of the study team at the largest community-based youth drop-in center, Family Health Options Kenya (FHOK), in Eldoret, where the peers already provide mentorship to adolescents. We will use the REAIM Framework to assess the reach, effectiveness, adoption, implementation, and maintenance of this intervention.

DETAILED DESCRIPTION:
Study Design The investigators will conduct a mixed-methods evaluation with peer providers, participants, and key delivery stakeholders such as FHOK staff. The investigators will collect quantitative data from: (1) peer mentors prior to their training and during the delivery of screening and treatment, (2) participants prior to entering treatment and after treatment. The investigators will track rates of retention, engagement, and attrition during screening and treatment delivery. Lastly, he investigators will collect qualitative data including interviews with 10 purposively sampled participants and Focus Groups with peer mentors and key delivery stakeholders post-treatment.

Study Sample. Based on available rates the investigators anticipate identifying around 360 teens with mental health problems in a 6-month period (20 teens per day, global rate of adolescent mental health problem ~15%)22. Linkage and treatment retention rates are low for this population ranging from 28%-78%23 . The investigators conservatively anticipate 45% attrition, resulting in a final sample of 162 receiving treatment. To estimate a pilot treatment effect for participants, a sample of 40 participants is needed to detect a small to medium treatment effect at 80% power and an alpha of 0.05. This effect is commensurate with those shown in previous RCT trials of PST delivered by lay providers24. As such, the investigators believe they will have enough participants to estimate a treatment effect and determine sample size estimates for a future cluster RCT trial. A power calculator was used to estimate a sample size needed to detect a medium effect size with a one group sample (Rosner B. Fundamentals of Biostatistics. 7th ed. Boston, MA: Brooks/Cole; 2011.) Notably, the effects in this study are preliminary indicators of implementation of the intervention and will be used to estimate power for a future, larger trial of PST.

The investigators will use convenience sampling, screening participants who present to the family health center for services. Such an approach best mirrors real world practice and can help provide key preliminary data around reach and service penetration to inform what implementation strategies may need to be applied later to improve implementation outcomes. Sample gender distribution will most likely mirror rates of gender distribution among youth attending Family Health services.

Data Collection Peer Logbooks/Forms: Peers will be provided screening and therapy logbooks to record all study data. These will be used to record number screened, screening results, and attendance to PST sessions for evaluating above metrics for reach, adoption, and implementation. Forms for SDQ, YTP, PHQ-9, and GAD-7 will be provided to peers for baseline screening, 1-month follow-up and 6-month follow-up for measuring effectiveness. Study Protocol will be for all logbooks and forms to be submitted to study office on a daily basis to be locked in a cabinet for confidentiality. The Youth Top Problem (YTP) assessment is a brief idiographic instrument designed to help identify and monitor youth problems that are especially important from the perspectives of the youth and the caregiver11, The Strengths and Difficulties Questionnaire (SDQ) a tool that assesses mental health problems among youth ( emotional symptoms, conduct problems ,Hyperactivity/inattention , peer relationship problems. social behavior) both of which have been used previously in Kenya,33. The investigators shall also use Patient Health Questionnaire (PHQ-9) a brief screening tool for depression. It is a 9-item self-report instrument for screening, and assessing the severity of depression, and examines for symptoms over the past two-week period. Each of the 9 items is rated as follows: 0 - "not at all", 1 - "Several days", 2 - "More than half the days", 3 - "Nearly every day". Interpretation of the total scores is as follows; 0-4 minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression50. The PHQ-9 has been validated in a low income Sub-Saharan Africa setting49. The investigators will use Generalized Anxiety Disorder 7 ( GAD-7 ) a tool for assessing generalized anxiety disorder, and these too have been widely used in the Kenyan setting. It is a seven item self-report instrument that examines for symptoms over the past two-week period. Each item is rated on a 4-point scale as follows: 0 - "not at all", 1 - "Several days", 2 - "More than half the days", 3 - "Nearly every day". Such scores have been shown to have a sensitivity of 89% and a specificity of 82%.51. The GAD-7 has been validated in a low income Sub-Saharan Africa setting49.

Written tests and Peer role plays: Peer mentor PST knowledge and competency will be measured with a written test assessing PST content and coded role plays (pre-post training) on clinical competency measured with the Enhancing Assessment of Common Therapeutic factors (ENACT) rating scale. This was previously used in Kenya to assess lay provider competency.26,27 Recording of PST sessions: PST sessions will be recorded to assess fidelity to PST measured with an adherence checklist outlining the steps of PST in each session (coding and analysis described below).

Study Procedures Community-Engaged Approach. This project will be guided by the principles of community-based participatory research in order to engage community stakeholders throughout study18. Such an approach helps to improve the quality, impact, and eventual sustainability of clinical treatment 19. Aligned with this approach, the project was developed due to the mental health needs described by FHOK. The proposed research will be guided by community partners including FHOK leadership, adolescents, MTRH representatives, and collaboration with Pamoja Mtaani, a youth group who mobilize youth to come to the drop-in center. The investigators will work with stakeholders to guide mobilization strategy and communications. Mobilizing the youth will be a key piece in ensuring the investigators meet the target sample size and understand reach. To get the desired number of adolescents to screen, the investigators shall incorporate activities that the youth have proposed.

Recruitment. The investigators will recruit FHOK peer-mentors aged 18-24 as providers and adolescents aged 12-18 years coming to the FHOK drop-in center as participants in this study. The peer mentors will require to have attained form 4 education and should have been volunteering with FHOK for a minimum of 6 months prior to recruitment. Out of 5 peer mentors, at least two will be from each gender

Peer-mentors/Providers. Peer mentors at FHOK are recruited from the community based on interest and willingness to volunteer time. On starting at FHOK, the peer mentors receive a one-week training on youth friendly services, peer-to-peer engagements and value clarification. The investigators will encourage all FHOK peers aged 18-24 who are not in school to apply to be peers for this study via flyers, text messages, presentations about the study, and word of mouth. Applications will consist of an initial application and interview process selecting 8-10 peers to attend the PST training with compensation provided for that time. After the training, post-training quiz results and role-plays will be used to select the five most qualified peer mentors to deliver the intervention with consent and research ethics training being provided after final selection.

Participants. For eligible adolescents, peer mentors will explain the study. If adolescents agree to participate, written assent will be obtained by the peer mentor and verbal phone consent for the parent/guardian. Youth will be eligible for screening if they are aged 12-18 years and reside within 30 minutes travel to the FHOK center. After screening, they will be eligible for treatment if they report elevated levels of mental health problems and are likely to remain in Eldoret for the duration of treatment. (If they will not remain in Eldoret, the investigators will try to assist them in linkage to other care.) The investigators will screen using the Swahili-language version of the Strengths and Difficulties Questionnaire (SDQ), the PHQ-9, and the GAD-7.

Treatment: Problem Solving Therapy (PST) The investigators will apply evidence-based Problem Solving Therapy (PST), a transdiagnostic, low-intensity approach shown to improve mental health problems among adolescents with demonstrated effectiveness in global settings20 21. PST for adolescents is a brief 5 session individual treatment with demonstrated efficacy when delivered by lay providers.32 PST is theorized to function by increasing adolescent capacity to cope with perceived and experienced stress through the use of problem- and emotion- focused coping skills that then allow engagement in positive, healthy activities. PST uses a straightforward approach amenable to use in new settings given its focus on idiographic problems, therefore session content is driven by the adolescent's presenting problem causing the most distress or impairment. The investigators will use the standardized, core steps of PST and existing manualized protocols including from the Friendship Bench study and the WHO protocol for Problem Management Plus.21,45 The peers will deliver PST through 5 structured counseling sessions of 30-60 minutes over a 4-6 week period. There are 5 core components of PST which including problem listing and identification, problem exploration, developing an action plan, implementation, and follow up.21 The components will be introduced in the first session and be reviewed in an iterative process across the session to help participants use this model for different problems.

Peer Mentor Training and Supervision To train and supervise peer mentors, the investigators will employ previously used approaches that have shown promising results in global mental health work.46 Further these procedures are open to iterative and collaborative refinements based on key delivery stakeholder (e.g., FHOK leadership, mentors) feedback as is a best practice in pilot studies. A 5-day training in screening for mental health problems and delivering PST, followed by 4 mock cases, and 2-observed cases prior to supervised practice. Observed sessions will serve as an opportunity of the on-site clinician to assess the peer-providers readiness to conduct a case with supervision.

Supervision. Peer-mentors will meet in groups led by a trained Psychologist to discuss cases, common challenges, and successes. As a first step, the investigators will take a tapered approach to supervision with higher intensity supervision at the start of implementation and reduced intensity over time. Across implementation, the peer- mentor groups will meet weekly. In month 1 of supervision, each group will be led by the trained psychologist. In month 2, the psychologist will lead the group bi-weekly, and two peer mentors, chosen by the larger group of peer-mentors, leading remaining meetings with psychologist support by phone if needed. In month 3 and beyond, the group will be led by two peer-mentors each week with psychologist support and consultation by phone as needed; every 6 weeks the psychologist will sit in on peer groups. For any emergencies or urgent questions, the psychologist will be available for consultation by phone.

ELIGIBILITY:
Inclusion Criteria:

* Meet any ONE of the following FOUR criteria: (1) a score a 5 or higher on the PHQ-9 OR (2) a score a 5 or higher on the GAD-7. Youth reporting suicidality on the PHQ-9 will be referred for mental health care and offered to enroll in PST.

Exclusion Criteria:

* intoxicated from any substance
* require urgent medical care
* receiving another mental health intervention
* show visible language difficulties (unable to understand assent process)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | On enrollment, at end of PST and six month follow-up
  This is a brief behavioral screening questionnaire for 2-17 year olds to assess mental health problems ( emotional symptoms, conduct problems, hyperactivity/inattention , peer relationship problems. social behavior). The overall SDQ score ranges from 0 to 50, with a higher score indicating abnormal behaviors.
Patient Health Questionnaire 9 (PHQ-9) | On enrollment, at end of PST and six month follow-up
  This is a brief screening tool for depression. Scale is from 0 to 27 with a higher score being more severe disease.
Generalized Anxiety Disorder 7 (GAD-7) | On enrollment, at end of PST and six month follow-up
  This is a tool for assessing generalized anxiety disorder. Scale is from 0 to 21 with a higher score being more severe disease.
Youth Top Problem (YTP) | On enrollment, at end of PST and six month follow-up
  a brief idiographic instrument designed to help identify and monitor youth problems that are especially important from the perspectives of the youth and the caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Turissini, MD, Principal Investigator — Indiana University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Uasin Gishu County, Kenya

IPD SHARING:
Plan to Share IPD: No